CLINICAL TRIAL: NCT00605046
Title: Evaluation of [123I] AV151 and SPECT as a Marker of Beta-amyloid Protein Deposition in Subjects With Alzheimer Disease (AD) in Comparison to Healthy Subjects
Brief Title: Evaluation of [123I] AV151 and SPECT in Subjects w/ AD in Comparison to Healthy Subjects
Acronym: AV151
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Scans showed no visual difference between affected subjects & healthy volunteers
Sponsor: Institute for Neurodegenerative Disorders (Other)
Responsible Party: Danna Jennings, MD, Institute for Neurodegenerative Disorders
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: AV151
Record Dates: First submitted 2008-01-16; First posted 2008-01-30 (Estimated); Last update posted 2010-10-06 (Estimated); Status verified 2010-10

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer; SPECT
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Asses [123I] AV151 and SPECT imaging (Experimental)
  Interventions: Drug: SPECT scan

INTERVENTIONS:
Drug: SPECT scan — AV151-01: Evaluation of [123I] AV151 and SPECT as a marker of beta-amyloid protein deposition in subjects with Alzheimer disease in comparison to healthy subjects

SUMMARY:
Purpose:

The main objectives of this proposal are as follows:

To assess the dynamic uptake and washout of 123-I AV151, a potential imaging biomarker for β-amyloid burden in brain, using single photon emission computed tomography (SPECT) in similarly aged healthy controls and Alzheimer's (AD) subjects

To perform blood metabolite characterization of 123-I AV151 in healthy and AD subjects to determine the metabolic fate and nature of metabolites in assessment of 123-I AV151 as a single photon computed tomography (SPECT) brain imaging agent

Evaluate the test/retest reproducibility of 123-I AV151 and SPECT in AD subjects and healthy controls

DETAILED DESCRIPTION:
General Design and Methods. The underlying goal of this study is to assess 123-I AV151 SPECT imaging as a tool to detect ß-amyloid deposition in the brain of AD research participants and age- and gender-matched healthy subjects. All study procedures will be conducted at the Institute for Neurodegenerative Disorders (IND) and Molecular NeuroImaging (MNI) in New Haven, CT. Approximately 20 patients with Alzheimers disease (AD) and 10 healthy controls will be recruited to participate in this study. Healthy controls will be examined to ensure that there is no evidence of neurodegenerative changes including cognitive decline. Informed consent will be obtained for all. All subjects will undergo a screening evaluation including baseline clinical laboratory testing, a baseline physical and neurological evaluation and baseline cognitive evaluations. Subjects will be asked to undergo a bolus injection of 123-I AV151. Subjects will undergo serial SPECT imaging scans and serial venous plasma sampling for measurement of 123-I AV151 in plasma (both protein bound and free) over a period of up to 6 hours. Subjects may be asked to undergo a second imaging visit between 2 and 6 weeks following the initial imaging visit following similar procedures to the initial imaging visit to evaluate the reproducibility of the imaging measure using this procedure. The imaging analyses will be performed by an image-processing specialist who will remain masked to the procedures employed with each imaging acquisition. The primary imaging outcome measure will be the brain regional distribution volumes expressed as a brain tissue to plasma ratio of the radioligand, 123-I AV151. Time to the peak uptake and amplitude of the peak uptake will be evaluated for all brain regions and the results for the AD patients and controls will be compared. For those subjects undergoing repeat imaging visits, the data from the initial scan will be compared to the second scan to determine which offers the reproducibility of the imaging outcome measure.

ELIGIBILITY:
INCLUSION CRITERIA: ALZHEIMER DISEASE

* The participant is 50 years or older.
* Written informed consent is obtained.
* Participants have a clinical diagnosis of Alzheimer's disease based on National Institute of Neurological and Communicative Disorders and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS/ADRDA) criteria.
* Mini-Mental Status Exam score < 25.
* Modified Hachinski Ischemia Scale score of ≤ 4.
* Geriatric Depression Scales (GDS) ≤ 10.
* For females, non-child bearing potential or negative urine or blood pregnancy test on day of 123-I AV151 injection.

EXCLUSION CRITERIA: ALZHEIMER DISEASE

* The subject has signs or symptoms of another neurodegenerative disease including Parkinson's disease, diffuse Lewy body dementia, or history of significant cerebrovascular disease.
* The subject has a clinically significant abnormal laboratory value and/or clinically significant unstable medical or psychiatric illness
* The subject has any disorder that may interfere with drug absorption distribution, metabolism, or excretion (including gastrointestinal surgery).
* The subject has evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, neurological, immunodeficiency, pulmonary, or other disorder or disease.
* Pregnancy

Concomitant therapy Patients may remain on a stable dose of anticholinesterase medication during the study. Use of donepezil (Aricept®), rivastigmine (Exelon®), galantamine (Razadyne®), tacrine (Cognex®), and memantine (Namenda®) are permitted during the study. Doses of these compounds must be stable for 2 months prior to the study. At each visit after the screening visit, the investigator will ask the patient whether any medications including OTC medications, were taken since the previous visit.

Use of antipsychotics for agitation and benzodiazepines for insomnia or anxiety is permitted. However, the use of these agents is not permitted within the 8 hours prior to administration of cognitive testing.

INCLUSION CRITERIA: HEALTHY VOLUNTEERS

* The participant is 50 years or older.
* Written informed consent is obtained.
* Negative history of neurological or psychiatric illness based on evaluation by a research physician.
* Mini-Mental Status Exam score ≥28.
* For females, non-child bearing potential or negative urine or blood pregnancy test on day of 123-I AV151 injection.

EXCLUSION CRITERIA: HEALTHY VOLUNEERS

* The subject has a clinically significant abnormal laboratory value and/or clinically significant unstable medical or psychiatric illness.
* The subject has any disorder that may interfere with drug absorption distribution, metabolism, or excretion (including gastrointestinal surgery).
* The subject has evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, neurological, immunodeficiency, pulmonary, or other disorder or disease.
* Pregnancy

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2007-08; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
AV151-01: Evaluation of [123I] AV151 and SPECT as a marker of beta-amyloid protein deposition in subjects with Alzheimer disease in comparison to healthy subjects | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Danna L Jennings, MD, Principal Investigator — Institute for Neurodegenerative Disorders
Locations (2):
- United States (2):
  - Institute for Neurodegenerative Disorders, New Haven, Connecticut
  - Molecular NeuroImaging, LLC, New Haven, Connecticut